CLINICAL TRIAL: NCT00253071
Title: Early Integrated Intervention in Severe Affective Disorders - a Randomized Controlled Trial.
Brief Title: Early Integrated Intervention in Severe Affective Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hovedstadens Sygehusfaelesskab (Other)
Collaborators: Rigshospitalet, Denmark (Other); Hvidovre University Hospital (Other); Amager Hospital (Other); Frederiksberg University Hospital (Other); Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Lars Vedel Kessing, Professor, MD, Hovedstadens Sygehusfaelesskab
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 31/04r
Record Dates: First submitted 2005-11-14; First posted 2005-11-15 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Depressive Disorder; Bipolar Disorder
Keywords: Prophylactic treatment; Pharmacological treatment; Psychological treatment
MeSH Terms: conditions — Depressive Disorder; Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A,2 (Active Comparator): Standard treatment: treatment as usual at a community psychiatric center, private psychiatrist or general practitioner.
  Interventions: Behavioral: Prophylactic combined medical and psychological treatment
- A, 1 (Experimental): Behavioral: Prophylactic combined medical and psychological treatment
  Medical treatment is naturalistic and evidence based according to international recommendations.
  Psychological treatment is either group psychoeducation or group cognitive behavioural therapy.
  Interventions: Behavioral: Prophylactic combined medical and psychological treatment

INTERVENTIONS:
Behavioral: Prophylactic combined medical and psychological treatment — Medical treatment is naturalistic and evidence based according to international recommendations.
  Psychological treatment is either group psychoeducation or group cognitive behavioural therapy.

SUMMARY:
The purpose of this study is to determine whether early integrated prophylactic combined medical and psychological outpatient treatment is associated with a better prognosis in patients with severe unipolar and bipolar affective disorders than standard treatment.

DETAILED DESCRIPTION:
Patients who have been hospitalised for unipolar or bipolar disorder have a poor prognosis with highly increased risk of recurrence of episodes and increased risk of psychosocial dysfunction. It seems as integrated prophylactic combined medical and psychological out-patient treatment may lead to a better long-term prognosis in patients with affective disorders in general. It has not been specifically investigated whether such integrated treatment may improve long-term outcome if the intervention is offered early in the course of the affective illness.

Subjects: Patients currently discharged from first, second or third hospitalisation ever from psychiatric department with a diagnosis of severe single depressive episode/recurrent depression or with a diagnosis of manic/mixed episode or bipolar disorder.

Comparison: Early intervention with integrated prophylactic combined medical and psychological outpatient treatment as offered by a clinic for affective disorders compared with standard outpatient treatment as offered by community psychiatric centres, private specialists in psychiatry or general practitioners.

ELIGIBILITY:
Inclusion Criteria:

1. Discharge diagnosis of severe single depressive episode, recurrent depression, manic/mixed episode or bipolar disorder

Exclusion Criteria:

1. Moderate to severe dementia
2. Incapable in understanding or reading danish
3. Earlier randomised to the trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 426 (Actual)
Dates: Start 2005-12; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Time to re-admission | 0-6 years

SECONDARY OUTCOMES:
Time to recurrence of an affective episode (depressive (MDI) or manic/mixed (MDQ)). | 1 and 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Lars V kessing, Professor, Principal Investigator — Department of psychiatry, University Hospital of Copenhagen, Denmark
Locations (1):
- Department of Psychiatry, University Hospital of Copenhagen, Denmark, Copenhagen, Denmark

REFERENCES:
- [Derived] Munkholm K, Kessing LV. Early specialised treatment for bipolar disorder: Long-term follow-up from the early intervention in affective disorders (EIA) randomised controlled trial. Acta Psychiatr Scand. 2024 Sep;150(3):138-147. doi: 10.1111/acps.13716. Epub 2024 Jun 2. PMID 38825333
- [Derived] Kessing LV, Hansen HV, Christensen EM, Dam H, Gluud C, Wetterslev J; Early Intervention Affective Disorders (EIA) Trial Group. Do young adults with bipolar disorder benefit from early intervention? J Affect Disord. 2014 Jan;152-154:403-8. doi: 10.1016/j.jad.2013.10.001. Epub 2013 Oct 10. PMID 24268595
- [Derived] Kessing LV, Hansen HV, Hvenegaard A, Christensen EM, Dam H, Gluud C, Wetterslev J; Early Intervention Affective Disorders (EIA) Trial Group. Treatment in a specialised out-patient mood disorder clinic v. standard out-patient treatment in the early course of bipolar disorder: randomised clinical trial. Br J Psychiatry. 2013 Mar;202(3):212-9. doi: 10.1192/bjp.bp.112.113548. Epub 2013 Jan 24. PMID 23349295
- [Derived] Hansen HV, Christensen EM, Dam H, Gluud C, Wetterslev J, Kessing LV; Early Intervention Affective Disorders (EIA) Trial Group. The effects of centralised and specialised intervention in the early course of severe unipolar depressive disorder: a randomised clinical trial. PLoS One. 2012;7(3):e32950. doi: 10.1371/journal.pone.0032950. Epub 2012 Mar 19. PMID 22442673
- [Derived] Kessing LV, Hansen HV, Christensen EM, Dam H, Gluud C, Wetterslev J; Early Intervention Affective Disorders (EIA) Group. The effects of centralised and specialised combined pharmacological and psychological intervention compared with decentralised and non-specialised treatment in the early course of severe unipolar and bipolar affective disorders--design of two randomised clinical trials. Trials. 2011 Feb 3;12:32. doi: 10.1186/1745-6215-12-32. PMID 21291564